CLINICAL TRIAL: NCT04572139
Title: Age-related Differences in the Response to a Combined Pituitary Stimulation Test With TRH, LHRH and ACTH
Brief Title: Age-related Differences in Response to Pituitary Stimulation Tests
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Riis, MD, Aalborg University Hospital
Other Study IDs: N-20200008
Record Dates: First submitted 2020-09-23; First posted 2020-10-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2023-08

CONDITIONS: Pituitary; Aging
MeSH Terms: conditions — Pituitary Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Young participants: 18-45 years old
  Interventions: Diagnostic Test: Pituitary stimulation test
- Old participants: 55-80 years old
  Interventions: Diagnostic Test: Pituitary stimulation test
- Oldest old participants: over 80 years old
  Interventions: Diagnostic Test: Pituitary stimulation test

INTERVENTIONS:
Diagnostic Test: Pituitary stimulation test — Pituitary stimulation with 0.1 mg LHRH, 0.2 mg TRH and 0.25 mg ACTH

SUMMARY:
The purpose of this study to age-related differences to the response of a combined pituitary stimulation test with TRH, LHRH and ACTH.

DETAILED DESCRIPTION:
Participants will be recruited in three different age intervals: 18-45 years, 55-80 years and 80+ years. These participants will all undergo the same stimulation test with 0.1 mg LHRH, 0.2 mg TRH, and 0.25 mg ACTH (Synachten). The tests will be perfomed at the same time of day for all particpants (between 08:15 and 08:45) and participants will be fasting for the test. Blood samples will be taken just before and at 10, 20, 30, 45, 60, 90 and 120 minutes following the stimulation test. Serum from blood samples will be stored at -20 degrees until analysis.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-45 or above 55.
* Healthy Volunteers

Exclusion Criteria:

* Medication or conditions affecting pituitary response (such as hormonal birth control, steriod use, thyroid disorders)
* Pregnancy or birth within the last year
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults across different age groups without conditions affecting pituitary function. Minimum sample size has been determined by power calculation to be 15 participants. The study aims to include up 24 particpants to increase power in the primary analysis.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Differences in area under the curve in TSH. | Immediately after procedure.
  Differences will be measured by calculating the area under the curve adjusted for the basal level for the time of the test period.
Differences in area under the curve in Prolactin. | Immediately after procedure.
  Differences will be measured by calculating the area under the curve adjusted for the basal level for the time of the test period.
Differences in area under the curve in LH. | Immediately after procedure.
  Differences will be measured by calculating the area under the curve adjusted for the basal level for the time of the test period.
Differences in area under the curve in FSH. | Immediately after procedure.
  Differences will be measured by calculating the area under the curve adjusted for the basal level for the time of the test period.
Differences in area under the curve in Cortisol. | Immediately after procedure.
  Differences will be measured by calculating the area under the curve adjusted for the basal level for the time of the test period.

OTHER OUTCOMES:
Differences in peak values in TSH | Immediately after procedure.
  Both absolute peak values and peak values relative to basal level will be calculated.
Differences in peak values in Prolactin | Immediately after procedure.
  Both absolute peak values and peak values relative to basal level will be calculated.
Differences in peak values in LH | Immediately after procedure.
  Both absolute peak values and peak values relative to basal level will be calculated.
Differences in peak values in FSH | Immediately after procedure.
  Both absolute peak values and peak values relative to basal level will be calculated.
Differences in peak values in Cortisol | Immediately after procedure.
  Both absolute peak values and peak values relative to basal level will be calculated.
Differences in time to peak for TSH. | Immediately after procedure.
  Delayed responses will be examined by inspecting curves and by comparing area under the curve at the different blood sampling time points during the test.
Differences in time to peak for Prolactin. | Immediately after procedure.
  Delayed responses will be examined by inspecting curves and by comparing area under the curve at the different blood sampling time points during the test.
Differences in time to peak for LH. | Immediately after procedure.
  Delayed responses will be examined by inspecting curves and by comparing area under the curve at the different blood sampling time points during the test.
Differences in time to peak for FSH. | Immediately after procedure.
  Delayed responses will be examined by inspecting curves and by comparing area under the curve at the different blood sampling time points during the test.
Differences in time to peak for Cortisol. | Immediately after procedure.
  Delayed responses will be examined by inspecting curves and by comparing area under the curve at the different blood sampling time points during the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Geriatric Medicine, Aalborg University Hospital, Aalborg, Northen Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No